CLINICAL TRIAL: NCT05419921
Title: Comparison of the Diagnostic Accuracy of Hysterosalpingo-lidocaine-foam Sonography Versus Hysterosalpingography in Tubal Patency Assessment to the Gold Standard of Laparoscopy and Dye Testing
Status: Terminated | Type: Observational
Why Stopped: The data collection team stopped recruiting cases.
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Tarek Elkhateb, Assistant lecturer, NewGiza University
Other Study IDs: IT28052022
Record Dates: First submitted 2022-06-08; First posted 2022-06-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Tubal Factor Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hysterosalpingo-lidocaine-foam-sonography combined with power doppler (HyLiFoSy-PD) — Women in the reproductive age group between 18- and 40-years old presenting with primary or secondary infertility who underwent HSG in the previous 5 years as a part of their infertility work-up with availability of good-quality HSG images, & did not get pregnant in this period, and gave no history of incidences that might affect their tubes, such as : abdominal surgery or laparoscopy, pelvic inflammatory disease, smoking, and intrauterine device insertion.
  Women fitting these inclusion criteria and scheduled for LDT as part of their infertility work up will be considered. HyLiFoSy-PD will be carried out few days before the already scheduled LDT.

SUMMARY:
This is a cross-sectional study that compares the diagnostic accuracy of Hysterosalpingo-lidocaine-foam sonography combined with power doppler (HyLiFoSy-PD) in the assessment of tubal patency, with the diagnostic accuracy of hysterosalpingogram (HSG), and to the gold standard of laparoscopy and dye testing.

ELIGIBILITY:
Inclusion Criteria:

1. Age group (18-40)
2. Informed signed Written consent.
3. Scheduled for LDT as a part of their infertility management
4. Have undergone HSG in the previous 5 years with the availability of good-quality HSG images.
5. No incident factors that might have affected the tubal status after she underwent HSG within the previous 5 years, such as ; abdominal surgery or laparoscopy, pelvic inflammatory disease, smoking, and intrauterine device insertion.

Exclusion Criteria:

1. LDT scheduled for a therapeutic purpose due to a known tubal or ovarian pathology
2. Lack of good-quality HSG images.
3. Withdrawal of consent.
4. Using contraception
5. Women outside reproductive age
6. Known allergy to lidocaine
7. Active pelvic inflammatory disease
8. Undiagnosed genital tract bleeding.
9. Evident tubal pathology (such as hydrosalpinx) or pregnancy diagnosed by transvaginal ultrasound (TV-US) prior to performing HyLiFoSy-PD 10- Incident factors that might have affected the tubal status after she underwent HSG within the previous 5 years, such as ; abdominal surgery or laparoscopy, pelvic inflammatory disease, smoking, and intrauterine device insertion.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women in the reproductive age group between 18- and 40-years old presenting with primary or secondary infertility who underwent HSG in the previous 5 years as a part of their infertility work-up with availability of good-quality HSG images, & did not get pregnant in this period, and gave no history of incidences that might affect their tubes, such as : abdominal surgery or laparoscopy, pelvic inflammatory disease, smoking, and intrauterine device insertion.
  Women fitting these inclusion criteria and scheduled for LDT as part of their infertility work up will be considered. HyLiFoSy-PD will be carried out few days before the already scheduled LDT.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of HyLiFoSy and HSG with reference to LDT, in terms of sensitivity, specificity, positive predictive value, negative predictive value, and overall accuracy. | July 2022- June 2024

SECONDARY OUTCOMES:
Evaluate the procedure associated pain | July 2022- June 2024
  Pain will be assessed during the procedure (after insertion of Foley's catheter, during injection of lidocaine-made gel foam) using the verbal rating scale (VRS). Interpretation will be like: no pain, mild pain, moderate pain, severe pain.
Evaluate the procedure duration | July 2022- June 2024
  Duration is calculated in minutes, from the introduction of Cusco speculum to the exit of Foley's catheter
Percentage of failed or inconclusive attempts and possible reasons for that | July 2022- June 2024
Incidence and rate of potential complications for example: vasovagal and allergic reactions, venous intravasation | July 2022- June 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Kasr Alainy OBGYN hospital, Cairo, AlQuahira, Egypt

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT05419921/Prot_SAP_000.pdf